CLINICAL TRIAL: NCT05899426
Title: Motor Learning-based Clinical Pilates Rehabilitation Protocol for Patients with Parkinson's Disease, Called @parkinsonpilates: Randomised Controlled Trial
Brief Title: Motor Learning-based Clinical Pilates Rehabilitation Protocol for Patients with Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Lefke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAYEK022.05
Record Dates: First submitted 2023-05-28; First posted 2023-06-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 2 groups will receive different exercise program for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor learning based clinical pilates (Experimental): Participants in this group will receive training for 60 minutes 2 times a week for 12 weeks and will be followed up with the same assessments at the 3rd months after the treatment.
  Interventions: Other: motor learning based clinical pilates
- Conventional Physiotherapy (Active Comparator): Participants in this group will receive training for 60 minutes 2 times a week for 12 weeks and will be followed up with the same assessments at the 3rd months after the treatment.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: motor learning based clinical pilates — The exercises will be created as function and goal. At least one stimulus will be given during each exercise (visual, tactile, auditory or vestibular). 2 different levels were determined for 3 months of treatment, according to the months. As the level increased, the intensity of the exercise increased. In general, the exercise intensity was increased according to the against gravity and the decreasing in the support area.
  Other Names: Parkinsonpilates
  Arms: Motor learning based clinical pilates
Other: Conventional Physiotherapy — This exercise program will include strengthening, stretching, posture exercises, balance and gait exercises. Aim is to improve muscle strength and prevent shortness of muscles. Also, balance and gait exercise aim to improve walking capacity.
  Other Names: Control group
  Arms: Conventional Physiotherapy

SUMMARY:
Individuals with Parkinson's disease demonstrate impaired motor learning, including a slower acquisition rate and poor retention, which may result from deficits in cognitive function, especially executive function. Considering the reduced motor learning ability in this patient group, exercises should be designed with a focus on strengthening sensory inputs and basic functional training. Therefore, the investigators established this program according to previous experience published study [NCT04063605]. Therefore, the feasibility of this rehabilitation protocol, which combines motor learning and clinical pilates principles and is adapted to the needs of individuals with Parkinson's disease, will be examined.

DETAILED DESCRIPTION:
The patients with Parkinson's Disease will be randomly assigned into two groups: Motor Learning based Clinical Pilates (MLCP) Group and Conventional Physiotherapy (CP) Group. Both groups will be treated for 12 weeks. The evaluation of the patients will be done before the beginning of exercise program, midterm evaluation in the 6th week and will be repeated at the end. Also there will be followed up evaluation with the same assessments at the 3rd month. Physical function/motor function of patients will be evaluated with The Unified Parkinson's Disease Rating Scale (UPDRS) III subscale, dynamic balance with Functional Reach Test (FRT), postural control and dynamic balance will also be evaluated with Berg Balance Scale and functional mobility by Timed Up and Go Test. Gait, balance and functional domains of the patients will be evaluated with Gait and Balance Scale (GABS), Nelson foot reaction test will be used for the reaction time.

ELIGIBILITY:
Inclusion Criteria:

* Having modified Hoehn & Yahr Scale grade 2-3 symptoms
* Be over 45 years old
* Having a score of 24 or 24< on the Mini Mental test
* To be able to read and write in Turkish
* Having at least 2 years Parkinson's Disease

Exclusion Criteria:

* Serious mental and psychological disorder
* Significant musculoskeletal disorders
* Lower extremity deformation
* Having another neurological disease
* Drug or dose change during treatment

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Nelson Foot Reaction Test | 5 minutes
  This test is measured using a ruler and this gives the simple reaction time. The participant sits against the wall with the toe at a distance of 2.5 cm and the heel at a distance of 5 cm from the wall. The test administrator holds the reaction ruler between the wall and the participant's foot and releases the ruler as soon as the participant is ready. The participant tries to hold the falling ruler by squeezing it against the wall. It will be measured 20 times. Five best and five worst values will be discarded and the average of the remaining measurement will be taken.
Gait and Balance Scale (Untimed Tasks) | 15 minutes
  Gait and Balance Scale (GABS) consists of historical information and examination of 14 different gait and balance parameters designed to assess the severity of these functional domains. Thirty-five patients with Parkinson's disease (PD), Hoehn and Yahr stages 1 - 3, were tested. Items 1 to 17 GABS are scored on a scale of 0 to 4 (0 being normal and 4 being the worst). Items 18- 24 are scored on a scale 0 to 1 or 0 to 2 (0 being normal and 1 or 2 being abnormal).
Gait and Balance Scale (Timed Tasks - Cadence) | 2 minutes
  Gait and Balance Scale (GABS) consists of timed tasks to assess gait speed and the 'up-and-go' test. Timed tasks provide valuable information about the gait cycle by measuring speed of walking, variation between the normal and fast gait speed, stand-walk-sit time and cadence.

SECONDARY OUTCOMES:
Functional reach test | 5 minutes
  A balance test designed to measure stability limits. The patient is asked to raise the dominant arm 90 ° and place it at the shoulder level and extend as far as it can go forward, without loss of movement or balance in the feet. Reduced ability to reach indicates an increased risk of falling in the future.
Timed-up and Go test | 5 minutes
  When the command is given, the patient gets up from a normal chair, walks 3 meters, turns and walks back to the chair and sits down. The time starts when the command is given and ends when the person sits back in the chair.
Berg Balance Scale | 15 minutes
  This test is used to measure a person&amp;amp;#39;s static and dynamic balance performance. It is effective in assessing postural control and predicting the risk of falling. It is a 14-item test that uses 0 to 4 sequential scoring for each item. The total score range is from 0 to 56 and a higher score indicates a better balance.
The Unified Parkinson&amp;amp;#39;s Disease Rating Scale (UPDRS) III. Subscale | 15 minutes
  The severity of motor symptoms will be assessed with the UPDRS III. (1) bradykinesia (finger taps, hand movements, rapid alternating movements of hand, leg agility, body bradykinesia and hypokinesia); (2) rigidity; (3) tremor (tremor at rest, action or postural tremor of hands); and (4) axial symptoms (arising from chair, posture, gait, postural stability).

CONTACTS AND LOCATIONS:
Overall Officials: Beliz Belgen Kaygısız, PT, PhD, Principal Investigator — European University of Lefke; Fahriye Çoban, PT, MSc, Principal Investigator — European University of Lefke
Locations (1):
- European University of Lefke, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No